CLINICAL TRIAL: NCT00704561
Title: Prospective, Randomized, Controlled Arm Study Comparing the Coverage of the Zotarolimus-eluting Stent vs Bare Metal Stent Implanted in ST- Elevation Myocardial Infarction (STEMI).
Brief Title: Vessel Wall Response of the Zotarolimus Drug-eluting Stent Implanted in AMI Assessed by Optical Coherence Tomography
Acronym: OCTAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Case Western Reserve University (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Giulio Guagliumi, Interventional cardiologist, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 457/2008
Record Dates: First submitted 2008-06-24; First posted 2008-06-25 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; Percutaneous Coronary Interventions; Optical Coherence Tomography; Thrombus
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DES - Zotarolimus Drug eluting stents (Active Comparator): Zotarolimus Drug eluting stents in overlap
  Interventions: Device: ENDEAVOR® drug-eluting stent (Medtronic, Santa Rosa, CA); Device: Coronary stent implantation
- BMS -Bare metal stent (Active Comparator): Bare metal stent
  Interventions: Device: DRIVER bare metal stent (Medtronic, Santa Rosa, Ca); Device: Bare Metal Coronary Stent

INTERVENTIONS:
Device: ENDEAVOR® drug-eluting stent (Medtronic, Santa Rosa, CA) — ENDEAVOR® drug-eluting stent implanted in acute myocardial infarction
  Arms: DES - Zotarolimus Drug eluting stents
Device: DRIVER bare metal stent (Medtronic, Santa Rosa, Ca) — DRIVER bare metal stent implanted in acute myocardial infarction
  Arms: BMS -Bare metal stent
Device: Coronary stent implantation — Comparison of Drug Eluting versus Bare Metal Stent
  Other Names: Zotarolimus Eluting Coronary Stent
  Arms: DES - Zotarolimus Drug eluting stents
Device: Bare Metal Coronary Stent — Comaprison between Drug Eluting and Bare Metal Coronary Stents
  Other Names: Driver Coronary Stent
  Arms: BMS -Bare metal stent

SUMMARY:
The objective of this study is to evaluate the completeness of struts coverage and vessel wall response (strut malapposition, neointima disomogeneities in texture) to the ENDEAVOR drug-eluting stent vs the DRIVER stent (bare metal stent of identical metallic platform) implanted for the treatment of the culprit lesion in ST-elevation acute myocardial infarction (STEMI). To investigate the completeness of the coverage as well as the number of uncovered stent struts per section (embedded, uncovered, malapposed) and the neointima texture, high resolution (~ 10-15 µm axial) intracoronary optical coherence tomography (OCT)will be used.

DETAILED DESCRIPTION:
Major concerns have been raised with regard to the safety of drug-eluting stents (DES) in patients with ST-elevation acute myocardial infarction (STEMI). Data from registry studies have suggested that implantation of DES during primary PCI could be associated with an increased risk for stent thrombosis, probably due to delayed arterial healing. Unlike first generation DES, zotarolimus-eluting stents seems to be associated with complete and uniform neointimal coverage. The objective of this prospective study is to measure the completeness of strut coverage and vessel wall response to the ENDEAVOR zotarolimus-eluting stent vs the DRIVER stent (bare metal stent of identical metallic platform) implanted in STEMI patients. Optical Coherence Tomography (OCT) that detects smaller degrees of stent strut coverage more accurately than IVUS will be used at 6 months follow-up. Intravascular ultrasound (IVUS) will be performed as per normal practice at any index procedures and at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myocardial MI with ST segment Elevation, within 12 hours from symptoms onset
* Native coronary artery disease with >70% diameter stenosis (no prior stent implant, no prior brachytherapy)
* Vessel size in between 2.5 and 3.75 mm
* Signed patient informed consent

Exclusion Criteria:

* Lesions in coronary artery bypass grafts
* Significant left main disease
* Killip class IV
* Reecent major bleeding (6 months)
* Renal failure with creatinine value > 2.5 mg/dl
* Allergy to aspirin and or clopidogrel/ticlopidine
* Patient in anticoagulant therapy
* IMA due to a stent thrombosis
* No suitable anatomy for OCT scan: (only ostial location, very tortuous anatomy, very distal or large vessels [≥ 3.75 mm in diameter])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Non inferiority OCT Number of uncovered Stent struts for Endeavor drug eluting stent vs Driver BMSbare metal stent | 6 months
  Non inferiority

SECONDARY OUTCOMES:
number of well apposed stent struts without neointima | 6 months
  number of well apposed stent struts without neointima
number of malapposed stent struts without neointima | 6 months
  number of malapposed stent struts without neointima
number of sections with > 30% uncovered struts/total struts | 6 months
  number of sections with > 30% uncovered struts/total struts
Number of sections with incomplete strut apposition | 6 months
  Number of sections with incomplete strut apposition
Adjudicated MACE(Death, re-MI, TLR) rate at 30 days and 6 months (non inferiority) | 6 months
  Adjudicated MACE(Death, re-MI, TLR) rate at 30 days and 6 months (non inferiority)
In segment OCT neontimal volume | 6 months
  In segment OCT neontimal volume

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — Cardiovascular Department Ospedali Riuniti di Bergamo
Locations (1):
- Ospedali Riuniti di Bergamo, Bergamo, Italy

REFERENCES:
- [Background] Luscher TF, Steffel J, Eberli FR, Joner M, Nakazawa G, Tanner FC, Virmani R. Drug-eluting stent and coronary thrombosis: biological mechanisms and clinical implications. Circulation. 2007 Feb 27;115(8):1051-8. doi: 10.1161/CIRCULATIONAHA.106.675934. PMID 17325255
- [Background] Daemen J, Wenaweser P, Tsuchida K, Abrecht L, Vaina S, Morger C, Kukreja N, Juni P, Sianos G, Hellige G, van Domburg RT, Hess OM, Boersma E, Meier B, Windecker S, Serruys PW. Early and late coronary stent thrombosis of sirolimus-eluting and paclitaxel-eluting stents in routine clinical practice: data from a large two-institutional cohort study. Lancet. 2007 Feb 24;369(9562):667-78. doi: 10.1016/S0140-6736(07)60314-6. PMID 17321312
- [Background] Kindermann M, Adam O, Werner N, Bohm M. Clinical Trial Updates and Hotline Sessions presented at the European Society of Cardiology Congress 2007: (FINESSE, CARESS, OASIS 5, PRAGUE-8, OPTIMIST, GRACE, STEEPLE, SCAAR, STRATEGY, DANAMI-2, ExTRACT-TIMI-25, ISAR-REACT 2, ACUITY, ALOFT, 3CPO, PROSPECT, EVEREST, COACH, BENEFiT, MERLIN-TIMI 36, SEARCH-MI, ADVANCE, WENBIT, EUROASPIRE I-III, ARISE, getABI, RIO). Clin Res Cardiol. 2007 Nov;96(11):767-86. doi: 10.1007/s00392-0591-z. Epub 2007 Oct 25. PMID 17955157
- [Background] Kastrati A, Dibra A, Spaulding C, Laarman GJ, Menichelli M, Valgimigli M, Di Lorenzo E, Kaiser C, Tierala I, Mehilli J, Seyfarth M, Varenne O, Dirksen MT, Percoco G, Varricchio A, Pittl U, Syvanne M, Suttorp MJ, Violini R, Schomig A. Meta-analysis of randomized trials on drug-eluting stents vs. bare-metal stents in patients with acute myocardial infarction. Eur Heart J. 2007 Nov;28(22):2706-13. doi: 10.1093/eurheartj/ehm402. Epub 2007 Sep 27. PMID 17901079
- [Background] Joner M, Finn AV, Farb A, Mont EK, Kolodgie FD, Ladich E, Kutys R, Skorija K, Gold HK, Virmani R. Pathology of drug-eluting stents in humans: delayed healing and late thrombotic risk. J Am Coll Cardiol. 2006 Jul 4;48(1):193-202. doi: 10.1016/j.jacc.2006.03.042. Epub 2006 May 5. PMID 16814667
- [Background] Nakazawa G, Finn AV, John MC, Kolodgie FD, Virmani R. The significance of preclinical evaluation of sirolimus-, paclitaxel-, and zotarolimus-eluting stents. Am J Cardiol. 2007 Oct 22;100(8B):36M-44M. doi: 10.1016/j.amjcard.2007.08.020. PMID 17950831
- [Background] Fajadet J, Wijns W, Laarman GJ, Kuck KH, Ormiston J, Munzel T, Popma JJ, Fitzgerald PJ, Bonan R, Kuntz RE; ENDEAVOR II Investigators. Randomized, double-blind, multicenter study of the Endeavor zotarolimus-eluting phosphorylcholine-encapsulated stent for treatment of native coronary artery lesions: clinical and angiographic results of the ENDEAVOR II trial. Circulation. 2006 Aug 22;114(8):798-806. doi: 10.1161/CIRCULATIONAHA.105.591206. Epub 2006 Aug 14. PMID 16908773
- [Background] Matsumoto D, Shite J, Shinke T, Otake H, Tanino Y, Ogasawara D, Sawada T, Paredes OL, Hirata K, Yokoyama M. Neointimal coverage of sirolimus-eluting stents at 6-month follow-up: evaluated by optical coherence tomography. Eur Heart J. 2007 Apr;28(8):961-7. doi: 10.1093/eurheartj/ehl413. Epub 2006 Nov 29. PMID 17135281
- [Background] Yamaguchi T, Terashima M, Akasaka T, Hayashi T, Mizuno K, Muramatsu T, Nakamura M, Nakamura S, Saito S, Takano M, Takayama T, Yoshikawa J, Suzuki T. Safety and feasibility of an intravascular optical coherence tomography image wire system in the clinical setting. Am J Cardiol. 2008 Mar 1;101(5):562-7. doi: 10.1016/j.amjcard.2007.09.116. Epub 2008 Jan 10. PMID 18307999
- [Background] Pinto Slottow TL, Waksman R. Overview of the 2007 Food and Drug Administration Circulatory System Devices Panel meeting on the endeavor zotarolimus-eluting coronary stent. Circulation. 2008 Mar 25;117(12):1603-8. doi: 10.1161/CIRCULATIONAHA.107.752261. No abstract available. PMID 18362244
- [Derived] Guagliumi G, Sirbu V, Bezerra H, Biondi-Zoccai G, Fiocca L, Musumeci G, Matiashvili A, Lortkipanidze N, Tahara S, Valsecchi O, Costa M. Strut coverage and vessel wall response to zotarolimus-eluting and bare-metal stents implanted in patients with ST-segment elevation myocardial infarction: the OCTAMI (Optical Coherence Tomography in Acute Myocardial Infarction) Study. JACC Cardiovasc Interv. 2010 Jun;3(6):680-7. doi: 10.1016/j.jcin.2010.04.005. PMID 20630463